CLINICAL TRIAL: NCT04316338
Title: Intermittent Theta-Burst Stimulation to Target Irritability in Adults With ASD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lawrence Fung, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-41458
Record Dates: First submitted 2019-09-24; First posted 2020-03-20 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Open-label design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active intermittent theta-burst stimulation (iTBS) (Experimental): 6 weeks of iTBS delivered at 80% resting motor threshold will be delivered to personalized regions in the prefrontal cortex based on each individual's functional connectivity.
  Interventions: Device: Intermittent theta-burst stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent theta-burst stimulation (iTBS) — Non-invasive brain stimulation technique

SUMMARY:
This study aims to demonstrate the feasibility, tolerability, safety and preliminary efficacy of 6 weeks of fMRI-guided iTBS delivered to personalized regions of the prefrontal cortex (PFC) in adults with ASD in reducing irritability in adults with ASD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ASD or Asperger's based on DSM-5 criteria as confirmed by a qualified clinician (including Dr. Fung), and if necessary the administration of Autism Diagnostic Interview-Revised (ADI-R) and/or Autism Diagnostic Observation Schedule-Generic (ADOS-G)
2. Age 22 to 55.
3. Adults who are physically healthy.
4. No significant current psychosocial stressors per history.
5. Full scale IQ > 50.
6. ABC-I score of 18 or greater.
7. if the participant is taking medication, they must be stable on this medication regiment for at least 4 weeks prior to baseline and agree to stay on these medications for the duration of the trial

Exclusion Criteria:

(f) Pre-term birth (<34 weeks' gestation) (g) Low birth weight (<2000 g). (h) DSM-5 diagnosis of other severe psychiatric disorder such as bipolar disorder or schizophrenia.

(i) Current use of benzodiazepines. (j) Use of other medications that modulate the GABA(A) receptor within 4 weeks of scanning (8 weeks for fluoxetine).

(k) History of alcoholism or substance abuse. (l) Active medical problems such as unstable seizures, congenital heart disease, endocrine disorders.

(m) Significant sensory impairments such as blindness or deafness. (n) Contraindication for MRI. (o) Pregnancy. (p) evidence of genetic syndrome.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist-irritability subscale (ABC-I) | Change across time: Baseline minus immediately after final treatment
  A parent/caregiver/clinician completed checklist (58-item) with an irritability subscale (15-item). Each item has a maximum score of 3, meaning that the irritability subscale has a maximum score of 45 and minimum score of 0. Higher scores indicate higher levels of irritability.

SECONDARY OUTCOMES:
Irritability Questionnaire | Baseline, every week of treatment (1-6), immediately after treatment, one month after treatment.
  A 21-item self-report measure of irritability. Each item is rated on how often (Never=0 to Most of the time=4) and the intensity (Not at all=0, Very much so=4) at which they occur.
Self-injury questionnaire (SIQ) | Baseline, immediately after treatment, one month after treatment.
  Self-report measure of self-injury, maximum 60 questions but participants only answer relevant questions. Five types of self-injurious behaviors are checked: scratching, bruising, cutting, burning, and biting oneself. It will assess the taxonomic specifications of self-injurious behavior (SIB- (e.g., type, frequency, duration)), but also the affective antecedents and consequences as well as the functions of each type of SIB.
THE MODIFIED OVERT AGGRESSION SCALE (MOAS) | Baseline, immediately after treatment, one month after treatment.
  Clinician rated scale of aggression. 4 items rated from 0-4. Maximum score is 16 with higher scores indicating higher levels of aggression, used to evaluate and document the "frequency and severity" of aggressive episodes.
Difficulties in Emotion Regulation Scale | Baseline, immediately after treatment, one month after treatment.
  Self-report measure of emotion regulation, evaluating individuals' levels of difficulties in regulating emotions. 36-item questionnaires. Each question rated from 1-5. Maximum score is 180 with higher scores indicating greater difficulty in emotion regulation. The instrument presents 36 items on a 5-point Likert scale of frequency (from 1 = almost never, to 5 = almost always).
The Adult Autism Quotient (AQ) | Baseline, immediately after treatment, one month after treatment.
  50-item self-report measure of autistic traits. Each of 50 statements are rated from 'definitely disagree' to 'definitely agree'.
Repetitive Behavior Scale-Revised (RBS-R) | Baseline, immediately after treatment, one month after treatment.
  43-item clinician rated scale measuring repetitive behaviors associated with ASD. Each item is rated from 0 (behavior does not occur) to 3 (behavior is a severe problem)
Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline, immediately after treatment, one month after treatment.
  10-item clinician rated measure of depressive symptoms. Each item is rated on a scale of 1-6.
Functional connectivity between areas involved in negative emotion regulation | Baseline, immediately after treatment, one month after treatment.
  Functional magnetic resonance imaging (fMRI) will be used to measure functional connectivity between areas involved in emotion regulation, previously shown to be involved in irritability. Areas of interest include: ventromedial prefrontal cortex, the amygdala, dorsolateral prefrontal cortex, the striatum.
EEG recordings | Baseline, immediately after treatment, one month after treatment.
  Electroencephalography (EEG) will be used to measure brain activity and connectivity before and after treatment. Resting-state EEG (5 minutes) with eyes open and TMS-evoked potential recordings will be taken before and after treatment. We are particularly interested in measuring gamma band activity (>30Hz) in participants while at rest.
Magnetic resonance spectroscopy (MRS) | Baseline, immediately after treatment, one month after treatment.
  MRS will be used to measure GABA levels in two brain areas of interest (ventromedial prefrontal cortex and amygdala) before and after treatment.
Aberrant Behavior Checklist-irritability subscale (ABC-I) | Change across time: Baseline minus one month after treatment
  A parent/caregiver/clinician completed checklist (58-item) with an irritability subscale (15-item). Each item has a maximum score of 3, meaning that the irritability subscale has a maximum score of 45 and minimum score of 0. Higher scores indicate higher levels of irritability.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fung, MD, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No